CLINICAL TRIAL: NCT03188315
Title: Studies of Small DNA Virus Encoded Oncogenes in Viral Carcinogenesis Using Laboratory Model Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heba Momen kamel (Other)
Responsible Party: Sponsor-Investigator, Heba Momen kamel, assistant lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17200086
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: DNA Virus Infections
MeSH Terms: conditions — DNA Virus Infections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases (Experimental): HPV detection HPV Genotyping HPV Oncogenes and oncoproteins
  Interventions: Genetic: HPV oncogenes
- control (Active Comparator): HPV detection HPV Genotyping HPV Oncogenes and oncoproteins
  Interventions: Genetic: HPV oncogenes

INTERVENTIONS:
Genetic: HPV oncogenes — PCR and oncogenes detection

SUMMARY:
Cancer is a devastating disease, presenting an immense disease burden to affected individuals and their families as well as health care systems with 10.9 million new cases and 6.7 million deaths per year. Approximately 12% of human cancers worldwide are caused by oncoviruses infection with more than 80% of cases occurring in the developing world.

Tumor viruses can be classified into two groups based on their genetic material;

1. DNA tumor viruses:

   1. Small DNA tumor viruses (Papilloma viruses, Polyoma viruses and adenoviruses).
   2. Complex DNA tumor viruses (Herpes viruses and Hepatitis B viruses).
2. RNA tumor viruses ( Hepatitis C viruses and human T-cell leukemia virus "HTLV").

There are around 100 types of HPV, with different variations in their genetic and oncogenic potential [5]. Thus, HPV genotypes are divided into 2 groups based on their vulnerability; High risk HPV (HR-HPV) and low risk HPV (LR-HPV).

The HPV genome encodes several oncoproteins [5]. E6 and E7 are the main genes responsible for cell transformation mediated by HR-HPV, and they modulate the activities of cellular proteins that regulate the cell cycle. Thus, the presence of E6/E7 can be a specific marker for diagnosing precancerous lesions by HPV.

Knowledge of the etiology of virus-mediated carcinogenesis, the networking of pathways involved in the transition from infection to cancer and the risk factors associated with each type of cancer, all suggest prophylactic and therapeutic strategies that may reduce the risk of virus-mediated cancer.

DETAILED DESCRIPTION:
Study subjects:

1. Inclusion criteria:

   * Age: 18 - 65 years old.
   * Women who are positive for HPV diagnosed by routine screening. Women willing to participate in the study and sign an informed consent
2. Exclusion criteria:

   * Age extremes (less than 18 years old or more than 65 years old).
   * Immuno-comprised patients, patients under steroid therapy or chemotherapy, or patients with serious medical illness that could affect their immune system.
   * Unknown medical history.

   Study Groups:
   * Group 1 (Cases): Patients known to have Cancer cervix with any degree of malignancy (diagnosed by routine screening or any other diagnostic tests)
   * Group 2 (Controls): Women sharing the same inclusion and exclusion criteria, but not known to have Cancer cervix

   Aim of The Study:
   1. Studying the role of HPV as an example of small DNA viruses in cell transformation and carcinogenesis.
   2. Determining the most HPV genotypes associated with high risks of cancer cervix occurrence.
   3. Detection of the HPV oncogenes playing role cell transformation and malignancy.
   4. Studying the role of viral DNA integration in cellular transformation and carcinogenesis.

      Study methods:

      Samples collection and storing:

      • Samples will be obtained from the cervix with the brush or swab\ by following the instructions corresponding to the type of collecting device.

      • Collection tubes will be stored at room temperature (15-30 °C).
      * Samples will be sent to the laboratory in less than 14 days following collection
      * The tubes can be preserved for 2-3 weeks at room temperature.

      HPV detection:
      * HPV cannot be propagated in tissue culture, and therefore, in most cases its accurate identification relies on molecular biology techniques, such as polymerase chain reaction (PCR).

      HPV Genotyping:

      • PCR-RFLP shows good discriminatory power by differentiating between HR and LR HPV genotypes, and it is possible to identify single or multiple infections .

      • In this technique, the amplified DNA is digested by restriction enzymes, resulting in DNA fragments of various lengths. Each fragment length is characteristic of a certain HPV genotype.

      • The commonest restriction enzymes are BamHI, Dd6eI, HaeIII, HinfI, PstI and RsaI.

      HPV Oncogenes and oncoproteins:

      • The main techniques used to detect mRNA for E6/E7 oncogenes are two commercial assays: PreTectW Proofer and APTIMAW HPV Assay. These techniques are based on transcription-mediated amplification of full-length E6/E7 transcripts using PCR.

      Statistical analysis:

      • Data will be analyzed by one-way analysis of variance using SPSS software version 24.0. Values will be expressed as mean ± S.D. For comparison between 2 groups, Student's t test will be used to determine whether the cases was significantly different from the control. Differences will be considered statistically significant at P<0.05, while P<0.01 will represent more significant change.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years old.
* Women who are positive for HPV diagnosed by routine screening.
* Women willing to participate in the study and sign an informed consent

Exclusion Criteria:

* Age extremes (less than 18 years old or more than 65 years old).
* Immuno-comprised patients, patients under steroid therapy or chemotherapy, or patients with serious medical illness that could affect their immune system.
* Unknown medical history.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
carcinogenesis | 6 months
  developing cancer cervix

IPD SHARING:
Plan to Share IPD: Undecided